CLINICAL TRIAL: NCT06624241
Title: Clinical Evaluation of Lipo-Curcumin Gel in Association with SRP for the Treatment of Stage III Periodontitis: a Randomized and Controlled Clinical Trial.
Brief Title: Effectiveness of SRP+ Lipo-curcumin Gel for the Treatment of Stage III Periodontitis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Michele Paolantonio, Head of Periodontology, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12062024
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-06

CONDITIONS: Periodontal Diseases; Periodontal Pocket; Periodontal Attachment Loss
Keywords: Curcumin; SRP; Liposome; Periodontitis
MeSH Terms: conditions — Periodontal Diseases; Periodontal Pocket; Periodontal Attachment Loss; Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Lipo-Curcumin gel + SRP (Experimental): After SRP the pocket defect will be filled with a Lipo-Curcumin gel and sealed with cyanoacrylate.
  Interventions: Procedure: Lipo-Curcumin gel + SRP
- Lipo gel + SRP (Active Comparator): After SRP the pocket defect will be filled with a Lipo gel and sealed with cyanoacrylate
  Interventions: Procedure: Lipo gel + SRP
- Discharged Gel + SRP (Active Comparator): After SRP the pocket defect will be filled with a discharged gel and sealed with cyanoacrylate
  Interventions: Procedure: Discharged Gel + SRP
- SRP alone (Active Comparator): SRP alone will be performed.
  Interventions: Procedure: SRP alone

INTERVENTIONS:
Procedure: Lipo-Curcumin gel + SRP — The pocket defect will be debrided with the use of fine ultrasonic tips and mini hand instruments and will be treated with the application of Lipo- Curcumin gel. The pocket will be sealed with cyanoacrylate.
  Arms: Lipo-Curcumin gel + SRP
Procedure: Lipo gel + SRP — The pocket defect will be debrided with the use of fine ultrasonic tips and mini hand instruments and will be treated with the application of Lipo gel. The pocket will be sealed with cyanoacrylate.
  Arms: Lipo gel + SRP
Procedure: Discharged Gel + SRP — The pocket defect will be debrided with the use of fine ultrasonic tips and mini hand instruments and will be treated with the application of discharged gel. The pocket will be sealed with cyanoacrylate.
  Arms: Discharged Gel + SRP
Procedure: SRP alone — The pocket defect will only be debrided with the use of fine ultrasound tips and mini hand instruments and no further treatment will be performed.
  Arms: SRP alone

SUMMARY:
The aim of the present study is to clinically and radiographically compare the effectivness of Scaling and Root Plannig (SRP) in association with lipo-curcumin gel (LC) respect SRP+ lipo-gel (L), SRP+ discharged (D) gel and SRP alone.

This study will be designed as a randomized clinical trial of 12-month duration. A total of 40 patients will be recruited and randomly equally distributed into 4 groups: an experimental group treated with SRP + LC, a first control group treated with SRP + L, a second control group treated with SRP+D and a third control group SRP alone.

Each defect will be treated with an ultrasonic scaler with dedicated thin tips for supra- and subgingival debridement associated with hand instrumentation under local anesthesia. Caution will be taken to preserve the stability of soft tissues. Following SRP, experimental and control sites will be randomly chosen. The test sites will be t filled with a Lipo-Curcumin gel and sealed with cyanoacrylate. In the first control group the defects will be be filled with a Lipo gel and sealed with cyanoacrylate. In the second control sites he pocket defect will be filled with a discharged gel and sealed with cyanoacrylate, in the third control group SRP alone will be performed.

Pre- and post-treatment clinical measurements were performed by an examiner blinded to the treatment modalities using a graded periodontal probe (HuFriedy UNC 15). Before the treatment and at 6 and 12 months post-treatment, all patients were examined by measuring the clinical attachment level, probing depth, gingival recession, full-mouth plaque score and bleeding on probing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of periodontitis stage III (grades A to C)
* on-smokers or former smokers who quit at least 1 year ago, and had not received any periodontal treatment in the 3 months prior to recruitment
* FMPS < 20% at baseline
* Furcation not involved
* Not Pregnant or Lactating
* Signed informed consent

Exclusion Criteria:

* Presence of uncontrolled systemic diseases that could affect treatment outcomes such as diabetes mellitus with an HbA1C>7%, rheumatoid arthritis or any form of immunosuppression
* Patients that had received systemic or local delivery of antibiotic therapy 6 weeks before enrollment
* Chronic intake of NSAIDs or steroids, currently

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Pocket Probing Depth (PPD) | 12 months
  Distance between the gingival margin and the bottom of the pocket.

SECONDARY OUTCOMES:
Clinical Attachment Level (CAL) | 12 months
  Distance between the CEJ and the bottom of the pocket
Gingival Recession (GR) | 12 months
  Distance between the CEJ and the gingival margin.
Full Mouth Plaque Score | 12 months
  Index that evaluates the general presence of bacterial plaque for all teeth. Through the passage of the probe, the presence of plaque deposits is reported for 4 surfaces for each tooth. A ratio is made between the contaminated surfaces and the total surfaces investigated to obtain a percentage value.
Full Mouth Bleeding Score | 12 months
  Index that evaluates the general presence of bleeding for all teeth. Through the insertion of a periodontal probe, the presence of bleeding on probing is signaled for 4 sites for each tooth. A ratio is made between the bleeding sites and the total sites investigated to obtain a percentage value.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Paolantonio, DDS, MD, Study Chair — University 'G. D'Annunzio' of Chieti
Locations (1):
- G. d'Annunzio University, Chieti, CH, Italy

IPD SHARING:
Plan to Share IPD: No